CLINICAL TRIAL: NCT02502266
Title: A Randomized Phase II/III Study of the Combination of Cediranib and Olaparib Compared to Cediranib or Olaparib Alone, or Standard of Care Chemotherapy in Women With Recurrent Platinum-Resistant or -Refractory Ovarian, Fallopian Tube, or Primary Peritoneal Cancer (COCOS)
Brief Title: Testing the Combination of Cediranib and Olaparib in Comparison to Each Drug Alone or Other Chemotherapy in Recurrent Platinum-Resistant Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Canadian Cancer Trials Group (Network); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-00651; NCI-2015-00651 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY005; s16-01681; NRG-GY005 (Other: NRG Oncology); NRG-GY005 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2015-07-17; First posted 2015-07-20 (Estimated); Results first posted 2025-05-06 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-07

CONDITIONS: Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Fallopian Tube Undifferentiated Carcinoma; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Adenocarcinoma; Ovarian Transitional Cell Carcinoma; Ovarian Undifferentiated Carcinoma; Primary Peritoneal Serous Adenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — cediranib; Magnetic Resonance Spectroscopy; olaparib; Paclitaxel; Taxes; liposomal doxorubicin; Doxorubicin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Phase II Arm I (reference regimen) (Active Comparator): Patients undergo physician's choice of standard of care chemotherapy, comprising either paclitaxel IV over 60 minutes on days 1, 8, 15, and 22 every 28 days (Regimen I); pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1 every 28 days (Regimen II); or topotecan hydrochloride IV over 30 minutes on days 1, 8, and 15 every 28 days or days 1-5 every 21 days (Regimen III). Treatment continues in the absence of disease progression or unacceptable toxicity. No modification of the assigned regimens, such as additional drugs (gemcitabine, or bevacizumab) is allowed. Patients also undergo CT and MRI throughout the study. (12/05/2016)
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Other: Questionnaire Administration; Drug: Topotecan; Drug: Topotecan Hydrochloride
- Phase II Arm II (cediranib maleate, olaparib) (Experimental): Patients receive cediranib maleate PO QD and olaparib PO BID. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout the study.
  Interventions: Drug: Cediranib; Drug: Cediranib Maleate; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib; Other: Questionnaire Administration
- Phase II Arm III (cediranib maleate) (Experimental): Patients receive cediranib maleate PO daily continuously. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout the study.
  Interventions: Drug: Cediranib; Drug: Cediranib Maleate; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration
- Phase II Arm IV (olaparib) (Experimental): Patients receive olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout the study. (In July 2018, the Data Monitoring Committee voted to exclude the olaparib alone regimen).
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib; Other: Questionnaire Administration
- Phase III Arm I (reference regimen) (Active Comparator): Patients undergo physician's choice standard of care chemotherapy as in Phase II Arm I. No modification of the assigned regimens, such as additional drugs (gemcitabine or bevacizumab) is allowed. Patients also undergo CT and MRI throughout the study. (12/05/2016)
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Other: Questionnaire Administration; Drug: Topotecan; Drug: Topotecan Hydrochloride
- Phase III Arm II (cediranib maleate, olaparib) (Experimental): Patients receive cediranib maleate PO and olaparib PO as in Phase II Arm II. Patients also undergo CT and MRI throughout the study.
  Interventions: Drug: Cediranib; Drug: Cediranib Maleate; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib; Other: Questionnaire Administration
- Phase III Arm III (single-agent cediranib maleate) (Experimental): Patients receive cediranib maleate PO as determined by the Phase II study. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout the study.
  Interventions: Drug: Cediranib; Drug: Cediranib Maleate; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Cediranib — Given PO
  Other Names: AZ-D2171; AZD 2171; AZD2171
  Arms: Phase II Arm II (cediranib maleate, olaparib); Phase II Arm III (cediranib maleate); Phase III Arm II (cediranib maleate, olaparib); Phase III Arm III (single-agent cediranib maleate)
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; AZD2171 Maleate; Recentin
  Arms: Phase II Arm II (cediranib maleate, olaparib); Phase II Arm III (cediranib maleate); Phase III Arm II (cediranib maleate, olaparib); Phase III Arm III (single-agent cediranib maleate)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
  Arms: Phase II Arm II (cediranib maleate, olaparib); Phase II Arm IV (olaparib); Phase III Arm II (cediranib maleate, olaparib)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Phase II Arm I (reference regimen); Phase III Arm I (reference regimen)
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; Dox-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; Pegylated Liposomal Doxorubicin; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
  Arms: Phase II Arm I (reference regimen); Phase III Arm I (reference regimen)
Other: Questionnaire Administration — Ancillary studies
Drug: Topotecan — Given IV
  Other Names: Hycamptamine; Topotecan Lactone
  Arms: Phase II Arm I (reference regimen); Phase III Arm I (reference regimen)
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Evotopin; Hycamptamine; Hycamtin; Nogitecan Hydrochloride; Potactasol; SKF S 104864 A; SKF S-104864-A; SKF S104864A; Topotec; Topotecan HCl; topotecan hydrochloride (oral)
  Arms: Phase II Arm I (reference regimen); Phase III Arm I (reference regimen)

SUMMARY:
This randomized phase II/III trial studies how well cediranib maleate and olaparib work when given together or separately, and compares them to standard chemotherapy in treating patients with ovarian, fallopian tube, or primary peritoneal cancer that has returned (recurrent) after receiving chemotherapy with drugs that contain platinum (platinum-resistant) or continued to grow while being treated with platinum-based chemotherapy drugs (platinum-refractory). Cediranib maleate and olaparib may stop the growth of tumor cells by blocking enzymes needed for cell growth. Chemotherapy drugs work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving cediranib maleate and olaparib together may cause more damage to cancer cells when compared to either drug alone or standard chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy and identify (in)active arm(s) of the combination of cediranib maleate (cediranib) and olaparib, cediranib alone, olaparib alone, and physician's choice standard of care chemotherapy, as measured by progression-free survival (PFS) in the setting of recurrent platinum-resistant or-refractory ovarian, primary peritoneal or fallopian tube cancer. (Phase II) II. To assess the efficacy of the combination of cediranib and olaparib, and cediranib monotherapy, as measured by overall survival (OS) and PFS, as compared to physician's choice standard of care chemotherapy in women with recurrent platinum-resistant or-refractory ovarian, primary peritoneal or fallopian tube cancer. (Phase III)

SECONDARY OBJECTIVES:

I. To assess the efficacy of the combination of cediranib and olaparib, cediranib alone, olaparib alone, and physician's choice standard of care chemotherapy, as measured by objective response rate (ORR: partial or complete response) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, in the setting of recurrent platinum-resistant or-refractory ovarian, primary peritoneal or fallopian tube cancer. (Phase II) II. To assess safety endpoints, as measured by frequency and severity of adverse events by Common Terminology Criteria for Adverse Events (CTCAE). (Phase II and Phase III) III. To assess the efficacy of the combination of cediranib and olaparib, and cediranib monotherapy, as measured by ORR as compared to physician's choice standard of care chemotherapy in the setting of recurrent platinum-resistant or-refractory ovarian, primary peritoneal or fallopian tube cancer. (Phase III)

OBJECTIVES WITH INTEGRATED BIOMARKERS:

I. To assess correlation of homologous recombination deficiency (HRD) status, as assessed via BROCA-HR assay with response, as measured by PFS and ORR. (Phase II) II. To evaluate the prognostic and predictive role of circulating endothelial cells (CEC) on comparative effectiveness of targeted therapies and reference chemotherapy. (Phase II) III. To evaluate quality of life data compliance, as measured by the 9-item Disease Related Symptoms (DRS-9) subscale of the National Comprehensive Cancer Network (NCCN)-Functional Assessment of Cancer Therapy (FACT) Ovarian Symptom Index (NFOSI) for utilization and analysis in the Phase III study. (Phase II) IV. To assess correlation of HRD status, as assessed via BROCA-HR assay with response, as measured by OS, PFS and ORR. (Phase III) V. To evaluate the prognostic and predictive role of circulating endothelial cells (CEC) on comparative effectiveness of targeted therapies and reference chemotherapy. (Phase III) VI. To assess the effect on disease-related symptoms (DRS) as measured by the 9-item DRS-P subscale of the NCCN-FACT Ovarian Symptom Index-18 (NFOSI-18), of single agent cediranib and cediranib/olaparib combination, compared to standard chemotherapy, in the setting of recurrent platinum-resistant or-refractory ovarian, primary peritoneal or fallopian tube cancer. (Phase III)

EXPLORATORY OBJECTIVES:

I. To assess exploratory biomarkers of potential HRD, including genomic scarring, BRCA1 methylation, BRCA1 protein expression, and mutations in NHEJ, and other genes that might modify HRD. (Phase II and Phase III) II. To evaluate the prognostic and predictive role of angiogenic biomarkers, as assessed by the Duke plasma angiome. (Phase II and Phase III) III. To assess the effect on secondary measures of quality of life, as assessed by the treatment side effects (TSE) and function/well-being (F/WB) subscales of the NFOSI-18, sensory neuropathy as measured by the FACT/GOG-Ntx-4, and health utility as measured by the EQ-5D, of single agent cediranib and cediranib/olaparib combination, compared to standard chemotherapy, in the setting of recurrent platinum-resistant or-refractory ovarian, primary peritoneal or fallopian tube cancer. (Phase III)

OUTLINE:

PHASE II: Patients are randomized to 1 of 4 treatment arms.

ARM I (REFERENCE REGIMEN): Patients undergo physician's choice of standard of care chemotherapy, comprising either paclitaxel intravenously (IV) over 60 minutes on days 1, 8, 15, and 22 every 28 days (Regimen I); pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1 every 28 days (Regimen II); or topotecan hydrochloride IV over 30 minutes on days 1, 8, and 15 every 28 days or days 1-5 every 21 days (Regimen III). Treatment continues in the absence of disease progression or unacceptable toxicity. No modification of the assigned regimens, such as additional drugs (gemcitabine, or bevacizumab) is allowed. Patients also undergo computed tomography (CT) and magnetic resonance imaging (MRI) throughout the study. (12/05/2016)

ARM II (CEDIRANIB MALEATE AND OLAPARIB): Patients receive cediranib maleate orally (PO) once daily (QD) and olaparib PO twice daily (BID). Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout the study.

ARM III (CEDIRANIB): Patients receive cediranib maleate PO daily continuously. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout the study.

ARM IV (OLAPARIB): Patients receive olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout the study. (In July 2018, the Data Monitoring Committee voted to exclude the olaparib alone regimen).

PHASE III: Patients are randomized to 1 of 3 treatment arms.

ARM I (REFERENCE REGIMEN): Patients undergo physician's choice standard of care chemotherapy as in Phase II Arm I. No modification of the assigned regimens, such as additional drugs (gemcitabine or bevacizumab) is allowed. Patients also undergo CT and MRI throughout the study. (12/05/2016)

ARM II (CEDIRANIB AND OLAPARIB): Patients receive cediranib maleate PO and olaparib PO as in Phase II Arm II. Patients also undergo CT and MRI throughout the study.

ARM III (SINGLE AGENT): Patients receive cediranib maleate PO as determined by the Phase II study. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed ovarian cancer, peritoneal cancer or fallopian tube cancer and must have a histological diagnosis of either serous or endometrioid cancer based on local histopathological findings; both endometrioid and serous histology should be high-grade for eligibility of non-mutation carriers; patients with clear cell, mixed epithelial, undifferentiated carcinoma, or transitional cell carcinoma histologies are also eligible, provided that the patient has a known deleterious germline BRCA1 or BRCA2 mutation identified through testing at a clinical laboratory

  * Note: Due to the long acceptance of BRCA testing through Myriad, Myriad testing will be accepted; if testing for BRCA is done by other organizations, documentation from a qualified medical professional (e.g., ovarian cancer specialty physician involved in the field, high risk genetics physician, genetics counselor) listing the mutation and confirming that the laboratory results showed a recognized germ line deleterious BRCA 1 or BRCA 2 mutation or BRCA rearrangement is required (12/05/2016); a copy of Myriad or other BRCA mutational analysis (positive or variants of unknown significance [VUS] or negative) reports will be requested but not required for study enrollment
* Patients should have recurrent platinum-resistant or- refractory disease - defined as disease that has progressed by imaging while receiving platinum or had recurrence within 6 months of the last receipt of platinum-based chemotherapy; rising CA125 only is not considered as platinum-resistant or refractory disease (12/05/2016)
* Phase II study: measurable disease by RECIST 1.1 criteria; if archival tumor sample is not available tumor sample from fresh biopsy is acceptable (12/05/2016)
* Phase III study: evaluable disease - defined as RECIST 1.1 measurable disease OR non-measurable disease (defined as solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions OR ascites and/or pleural effusion that has been pathologically demonstrated to be disease-related in the setting of a cancer antigen [CA]125 >= 2 x upper limit of normal [ULN])
* No more than 3 prior treatment regimens (including primary therapy; no more than 1 prior non-platinum based therapy in the platinum-resistant/-refractory setting); hormonal therapies used as single agents (i.e. tamoxifen, aromatase inhibitors) will not count towards this line limit (12/05/2016)
* Patients may not have had a prior anti-angiogenic agent in the recurrent setting; prior use of bevacizumab in the upfront or upfront maintenance setting is allowed
* Patients may not have previously received a PARP-inhibitor
* Patient must have provided study specific informed consent prior to study entry
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 or 2
* Absolute neutrophil count >= 1,500/mcL (12/05/2016)
* Platelets >= 100,000/mcL (12/05/2016)
* Hemoglobin >= 10 g/dL (12/05/2016)
* Total bilirubin within =< 1.5 times the upper limit of normal (ULN) institutional limits (12/05/2016)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN; if intrahepatic liver metastases are present, AST and ALT must be =< 5 times institutional ULN (12/05/2016)
* Creatinine =< 1.5 x the institutional ULN (12/05/2016)
* Urine protein: creatinine ratio urine protein creatinine (UPC) of =< 1 OR less than or equal to 2+ proteinuria on two consecutive dipsticks taken no less than 1 week apart; UPC is the preferred test; patients with 2+ proteinuria on dipstick must also have a 24-hour urine collection demonstrating protein of =< 500 mg over 24 hours (12/05/2016)
* Toxicities of prior therapy (excepting alopecia) should be resolved to less than or equal to grade 1 as per CTCAE; patients with long-standing stable grade 2 neuropathy may be considered after discussion with the study chair.
* Adequately controlled blood pressure (systolic blood pressure [SBP] =< 140; diastolic blood pressure [DBP] =< 90 mmHg) on maximum of three antihypertensive medications; patients must have a BP of =< 140/90 mmHg taken in the clinic setting by a medical professional within 2 weeks prior to starting study; it is strongly recommended that patients who are on three antihypertensive medications be followed by a cardiologist or a primary care physician for management of BP while on protocol; patients must be willing and able to check and record daily blood pressure readings; blood pressure cuffs will be provided to patients randomized to cediranib alone and the combination of olaparib and cediranib arms (12/05/2016)
* Adequately controlled thyroid function, with no symptoms of thyroid dysfunction and thyroid-stimulating hormone (TSH) within normal limits (12/05/2016)
* Able to swallow and retain oral medications and without gastrointestinal (GI) illnesses that would preclude absorption of cediranib or olaparib
* Age >= 18 years
* Cediranib has been shown to terminate fetal development in the rat, as expected for a process dependent on VEGF signaling; for this reason, women of child-bearing potential must have a negative pregnancy test prior to study entry; women of child-bearing potential must agree to use two reliable forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 weeks after cediranib discontinuation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Olaparib adversely affects embryofetal survival and development in the rat; for this reason, women of child-bearing potential must have a negative pregnancy test prior to study entry; women of child-bearing potential must agree to use must agree to use two reliable forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 3 months after the last dose of olaparib; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) of starting treatment or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; patients may not have had hormonal therapy within 2 weeks prior to entering the study; patients receiving raloxifene for bone health as per Food and Drug Administration (FDA) indication may remain on raloxifene absent other drug interactions (12/05/2016)
* Any other investigational agents within the past 4 weeks
* Prior treatment affecting the VEGF/VEGFR pathway or the angiopoietin pathway in the recurrent setting, including but not limited to thalidomide, bevacizumab, sunitinib, sorafenib, pazopanib, cediranib, nintedanib, and trebananib; bevacizumab used in the upfront setting in conjunction with chemotherapy and/or as maintenance to treat newly diagnosed disease will be allowed
* Prior use of PARP-inhibitors
* CA-125 only disease without Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 measurable or otherwise evaluable disease
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to starting cediranib
* Current signs and/or symptoms of bowel obstruction or signs and/or symptoms of bowel obstruction within 3 months prior to starting study drugs
* History of intra-abdominal abscess within the past 3 months
* History of gastrointestinal perforation; patients with a history of abdominal fistula will be considered eligible if the fistula was surgically repaired or has healed, there has been no evidence of fistula for at least 6 months, and patient is deemed to be at low risk of recurrent fistula (12/05/2016)
* Dependency on IV hydration or total parenteral nutrition (TPN)
* Any concomitant or prior invasive malignancies with the following curatively treated exceptions:

  * Treated limited stage basal cell or squamous cell carcinoma of the skin
  * Carcinoma in situ of the breast or cervix
  * Primary endometrial cancer meeting the following conditions: stage not greater than IA, grade 1 or 2, no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous/serous, clear cell, or other Federation of Gynecology and Obstetrics (FIGO) grade 3 lesions (12/05/2016)
  * Prior cancer treated with a curative intent with no evidence of recurrent disease 5 years following diagnosis and judged by the investigator to be at low risk of recurrence
* Patients with untreated brain metastases, spinal cord compression, or evidence of symptomatic brain metastases or leptomeningeal disease as noted on computed tomography (CT) or magnetic resonance imaging (MRI) scans should not be included on this study, since neurologic dysfunction may confound the evaluation of neurologic and other adverse events; patients with treated brain metastases and resolution of any associated symptoms must demonstrate stable post-therapeutic imaging for at least 6 months following therapy prior to starting study drug
* Patients with any of the following:

  * History of myocardial infarction within six months
  * Unstable angina
  * Resting electrocardiogram (ECG) with clinically significant abnormal findings
  * New York Heart Association functional classification of III or IV
* If cardiac function assessment is clinically indicated or performed: left ventricular ejection fraction (LVEF) less than normal per institutional guidelines, or < 55%, if threshold for normal not otherwise specified by institutional guidelines

  * Patients with the following risk factors should have a baseline cardiac function assessment:

    * Prior treatment with anthracyclines
    * Prior treatment with trastuzumab
    * Prior central thoracic radiation therapy (RT), including RT to the heart
    * History of myocardial infarction within 6 to 12 months (Patients with history of myocardial infarction within 6 months are excluded from the study)
    * Prior history of impaired cardiac function
* History of stroke or transient ischemic attack within six months
* Clinical significant peripheral vascular disease or vascular disease (aortic aneurysm or aortic dissection)
* Evidence of coagulopathy or bleeding diathesis; therapeutic anticoagulation for prior thromboembolic events is permitted
* Evidence suggestive of myelodysplastic syndrome (MDS) or acute myelogenous leukemia (AML) on peripheral blood smear or bone marrow biopsy, if clinically indicated

  * No prior allogeneic bone marrow transplant or double umbilical cord blood transplantation (dUBCT)
* Patients may not use any complementary or alternative medicines including natural herbal products or folk remedies as they may interfere with the effectiveness of the study treatments
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (other than atrial fibrillation with controlled ventricular rate), or psychiatric illness/social situations that would limit compliance with study requirements (12/05/2016)
* Known human immunodeficiency virus (HIV)-positive individuals are ineligible because of the potential for pharmacokinetic interactions with cediranib or olaparib; in addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy
* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible

  * Strong inhibitors and inducers of UGT/PgP should be used with caution (12/05/2016)
* Pregnant women are excluded from this study because cediranib and olaparib are agents with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with cediranib and olaparib, breastfeeding should be discontinued if the mother is treated with cediranib or olaparib; these potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2026-07-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-min Lee, Principal Investigator — NRG Oncology
Locations (398):
- United States (370):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Auburn Faith Hospital, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Marin Cancer Care Inc, Greenbrae, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - WellStar Health System Inc, Marietta, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - WellStar North Fulton Hospital, Roswell, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - WellStar Vinings Health Park, Smyrna, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - UChicago Medicine Comprehensive Cancer Center - Saint Joseph Hospital, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Associates In Womens Health, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Women's Cancer Care-Covington, Covington, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - TidalHealth Richard A Henson Cancer Institute, Ocean Pines, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Thompson Cancer Survival Center - West, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Intermountain Medical Center, Murray, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - Women's Cancer Center of Seattle, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Monongalia Hospital, Morgantown, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
- Canada (13):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Algoma District Cancer Program Sault Area Hospital, Sault Ste. Marie, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
- Japan (7):
  - Ehime University Hospital, Tōon, Ehime
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - The Cancer Institute Hospital Of JFCR, Koto-ku, Tokyo
  - Kindai University, Osaka
  - Saitama Medical University International Medical Center, Saitama
  - National Cancer Center Hospital, Tokyo
- Centro Comprensivo de Cancer de UPR, San Juan, Puerto Rico
- South Korea (7):
  - Keimyung University-Dongsan Medical Center, Dalseo-gu, Daegu
  - Seoul National University Bundang Hospital, Seongnam, Kyeonggi-do
  - Gachon University Gil Hospital, Incheon
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Korea Cancer Center Hospital, Seoul

REFERENCES:
- [Derived] Lee JM, Brady MF, Miller A, Moore RG, MacKay H, McNally L, Lea J, Street D, Lheureux S, McDonald ME, Duska LR, Cantuaria G, Kavecansky J, Leath CA 3rd, Powell M, Cadungog MG, Rose PG, Kim YM, Huang HQ, Provencher M, Wenzel LB, Bookman MA, Kohn EC, Secord AA. Cediranib and Olaparib Combination Compared With Cediranib or Olaparib Alone, or Chemotherapy in Platinum-Resistant or Primary Platinum-Refractory Ovarian Cancer: NRG-GY005. J Clin Oncol. 2024 Dec 20;42(36):4305-4316. doi: 10.1200/JCO.24.00683. Epub 2024 Oct 3. PMID 39361946

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study opened on 05 Feb 2016. Phase 2 accrual completed on 16 Jun 2017 with 213 patients randomly assigned to 4 treatment arms. Enrollment to Arm IV (olaparib) was suspended after DMC review and 52 patients on Arm IV during phase 2 not included in phase 3 analysis. Phase 3 accrual started on 17 Dec 2018 with 349 patients including 4 Japanese patients enrolled to Phase 3 three arms by 02 Oct 2020. After that, 20 Japanese patients were enrolled but not included in the phase 3 analysis.
Groups:
- Arm I (Reference Regimen): Patients undergo physician's choice of standard of care chemotherapy, comprising either paclitaxel IV over 60 minutes on days 1, 8, 15, and 22 every 28 days (Regimen I); pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1 every 28 days (Regimen II); or topotecan hydrochloride IV over 30 minutes on days 1, 8, and 15 every 28 days or days 1-5 every 21 days (Regimen III). Treatment continues in the absence of disease progression or unacceptable toxicity. No modification of the assigned regimens, such as additional drugs (gemcitabine, or bevacizumab) is allowed. Patients also undergo CT and MRI throughout the study. (12/05/2016)
  Computed Tomography: Undergo CT
  Magnetic Resonance Imaging: Undergo MRI
  Paclitaxel: Given IV
  Pegylated Liposomal Doxorubicin Hydrochloride: Given IV
  Questionnaire Administration: Ancillary studies
  Topotecan: Given IV
  Topotecan Hydrochloride: Given IV
- Arm II (Cediranib Maleate, Olaparib): Patients receive cediranib maleate PO QD and olaparib PO BID. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout the study.
  Cediranib: Given PO
  Cediranib Maleate: Given PO
  Computed Tomography: Undergo CT
  Magnetic Resonance Imaging: Undergo MRI
  Olaparib: Given PO
  Questionnaire Administration: Ancillary studies
- Arm III (Cediranib Maleate): Patients receive cediranib maleate PO daily continuously. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout the study.
  Cediranib: Given PO
  Cediranib Maleate: Given PO
  Computed Tomography: Undergo CT
  Magnetic Resonance Imaging: Undergo MRI
  Questionnaire Administration: Ancillary studies
- Arm IV (Olaparib) (Phase II Only): Patients receive olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout the study. (In July 2018, the Data Monitoring Committee voted to exclude the olaparib alone regimen).
  Computed Tomography: Undergo CT
  Magnetic Resonance Imaging: Undergo MRI
  Olaparib: Given PO
  Questionnaire Administration: Ancillary studies
- Arm V (Arm I Regimen: JP Patients Enrolled After P3 Cutoff): Patients undergo physician's choice of standard of care chemotherapy, comprising either paclitaxel intravenously (IV) over 60 minutes on days 1, 8, 15, and 22 every 28 days (Regimen I); pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1 every 28 days (Regimen II); or topotecan hydrochloride IV over 30 minutes on days 1, 8, and 15 every 28 days or days 1-5 every 21 days (Regimen III). Treatment continues in the absence of disease progression or unacceptable toxicity. No modification of the assigned regimens, such as additional drugs (gemcitabine, or bevacizumab) is allowed. Patients also undergo computed tomography (CT) and magnetic resonance imaging (MRI) throughout the study. (12/05/2016) Patients enrolled from Japan after the Phase III cutoff.
- Arm VI: (Arm II Regimen: JP Patients Enrolled After P3 Cutoff): Patients receive cediranib maleate orally (PO) once daily (QD) and olaparib PO twice daily (BID). Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout the study. Patients enrolled from Japan after the Phase III cutoff.
- Arm VII: (Arm III Regimen: JP Patients Enrolled After P3 Cutoff): Patients receive cediranib maleate PO daily continuously. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout the study. Patients enrolled from Japan after the Phase III cutoff.
Period: Overall Study
Arm/Group | Arm I (Reference Regimen) | Arm II (Cediranib Maleate, Olaparib) | Arm III (Cediranib Maleate) | Arm IV (Olaparib) (Phase II Only) | Arm V (Arm I Regimen: JP Patients Enrolled After P3 Cutoff) | Arm VI: (Arm II Regimen: JP Patients Enrolled After P3 Cutoff) | Arm VII: (Arm III Regimen: JP Patients Enrolled After P3 Cutoff)
Started | 173 | 167 | 170 | 52 | 5 | 8 | 7
Completed | 124 | 146 | 139 | 0 | 3 | 5 | 6
Not Completed | 49 | 21 | 31 | 52 | 2 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 30 | 15 | 16 | 0 | 0 | 0 | 0
Not completed — Still on Treatment | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other Reasons | 19 | 6 | 14 | 0 | 1 | 1 | 0
Not completed — Arm 4 Discontinued | 0 | 0 | 0 | 52 | 0 | 0 | 0
Not completed — Never treated | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized Subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Reference Regimen) | Arm II (Cediranib Maleate, Olaparib) | Arm III (Cediranib Maleate) | Arm IV (Olaparib) (Phase II Only) | Arm V (Arm I Regimen: JP Patients Enrolled After P3 Cutoff) | Arm VI: (Arm II Regimen: JP Patients Enrolled After P3 Cutoff) | Arm VII: (Arm III Regimen: JP Patients Enrolled After P3 Cutoff) | Total
Number analyzed (Participants) | 173 | 167 | 170 | 52 | 5 | 8 | 7 | 582
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 3
  30-39 years | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 5
  40-49 years | 9 | 14 | 14 | 4 | 1 | 1 | 1 | 44
  50-59 years | 41 | 34 | 36 | 13 | 1 | 2 | 2 | 129
  60-69 years | 63 | 60 | 72 | 22 | 0 | 3 | 3 | 223
  70-79 years | 48 | 48 | 45 | 11 | 3 | 2 | 1 | 158
  >= 80 years | 7 | 9 | 3 | 1 | 0 | 0 | 0 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 167 | 170 | 52 | 5 | 8 | 7 | 582
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 3 | 4 | 0 | 0 | 0 | 19
  Not Hispanic or Latino | 161 | 157 | 165 | 46 | 5 | 8 | 7 | 549
  Unknown or Not Reported | 6 | 4 | 2 | 2 | 0 | 0 | 0 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 6
  Asian | 19 | 12 | 11 | 0 | 5 | 8 | 7 | 62
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Black or African American | 11 | 6 | 11 | 4 | 0 | 0 | 0 | 32
  White | 135 | 142 | 142 | 45 | 0 | 0 | 0 | 464
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 5 | 3 | 1 | 0 | 0 | 0 | 16

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) (Phase II Only)
Description: Progression free survival (PFS) was defined as the number of months between study enrollment and documentation of disease progression (RECIST 1.1) or death from any cause. Patients still alive and disease free at the last follow-up were censored on the date of last CT Scan, or the CT Scan date prior to two missed assessments.
  Disease progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: The protocol required lesion assessments every 9 weeks from cycle 1, day 1 for the first year, then every 12 weeks thereafter until disease progression. Approximately 42 months.
Population: All subjects randomized at Phase II.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Reference Regimen) | Arm II (Cediranib Maleate, Olaparib) | Arm III (Cediranib Maleate) | Arm IV (Olaparib) (Phase II Only)
Number analyzed (Participants) | 53 | 55 | 53 | 52
Months | 2.3 [2.1 to 4.2] | 6.2 [3.9 to 8.2] | 3.4 [2.3 to 4.8] | 2.3 [2.0 to 2.8]
Statistical Analysis 1: Comparison: Arm I (Reference Regimen) vs Arm II (Cediranib Maleate, Olaparib); Experimental regimens with at least a 17% reduction in the estimated PFS event rate (compared to standard chemotherapy) (HR estimate < 0.83) were recommended for further evaluation in the phase III trial; Test type: Superiority; Hazard Ratio (HR) = 0.649, 95% CI 2-sided [0.424 to 0.995] — The hazard ratio estimate compares Cediranib and Olaparib to chemotherapy. If Cediranib and Olaparib is superior, the hazard ratio is <1.0
Statistical Analysis 2: Comparison: Arm I (Reference Regimen) vs Arm III (Cediranib Maleate); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Hazard Ratio (HR) = 0.832, 95% CI 2-sided [0.539 to 1.284] — The hazard ratio estimate compares Cediranib to chemotherapy. If Cediranib is superior, the hazard ratio is <1.0
Statistical Analysis 3: Comparison: Arm I (Reference Regimen) vs Arm IV (Olaparib) (Phase II Only); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Hazard Ratio (HR) = 1.149, 95% CI 2-sided [0.745 to 1.773] — The hazard ratio estimate compares Olaparib to chemotherapy. If Olaparib is superior, the hazard ratio is <1.0

2. Primary Outcome: Progression-free Survival (PFS) (Phase III Only)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All randomized subjects in Arms I - VII (excluding Arm IV).
  Arm 4 (Olaparib alone) was not continued in the Phase III part for its lack of efficacy after the completion of the Phase II portion. No further analyses were performed or reported for this arm.
  The primary endpoint analysis also did not include 20 Japanese patients who were enrolled after the primary Phase III endpoint was reached.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm V: (Arm 1 Regimen: JP Patients Enrolled After P3 Cutoff): Patients undergo physician's choice of standard of care chemotherapy, comprising either paclitaxel intravenously (IV) over 60 minutes on days 1, 8, 15, and 22 every 28 days (Regimen I); pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1 every 28 days (Regimen II); or topotecan hydrochloride IV over 30 minutes on days 1, 8, and 15 every 28 days or days 1-5 every 21 days (Regimen III). Treatment continues in the absence of disease progression or unacceptable toxicity. No modification of the assigned regimens, such as additional drugs (gemcitabine, or bevacizumab) is allowed. Patients also undergo computed tomography (CT) and magnetic resonance imaging (MRI) throughout the study. (12/05/2016) Patients enrolled from Japan after the Phase III cutoff.
Arm/Group | Arm I (Reference Regimen) | Arm II (Cediranib Maleate, Olaparib) | Arm III (Cediranib Maleate) | Arm V: (Arm 1 Regimen: JP Patients Enrolled After P3 Cutoff) | Arm VI: (Arm II Regimen: JP Patients Enrolled After P3 Cutoff) | Arm VII: (Arm III Regimen: JP Patients Enrolled After P3 Cutoff)
Number analyzed (Participants) | 173 | 167 | 170 | 5 | 8 | 7
months | 3.4 [2.4 to 4.3] | 5.2 [4.2 to 6.2] | 4.0 [3.2 to 4.3] | 4.2 [2.1 to NA] — The sample size is not sufficient for the estimation of the upper bound of the CI. | 5.3 [2.5 to 12.6] | 4.1 [2.3 to 4.8]
Statistical Analysis 1: Comparison: Arm I (Reference Regimen) vs Arm II (Cediranib Maleate, Olaparib); Arm IV was suspended for futility at the end of Phase 2 analysis, so was not analyzed at the final analysis; Test type: Superiority; p = 0.145, Log Rank — The log rank test was stratified by the factors provided at randomization; Hazard Ratio (HR) = 0.796, 98% CI 2-sided [0.597 to 1.060] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm I (Reference Regimen) vs Arm III (Cediranib Maleate); Arm IV was suspended for futility at the end of Phase 2 analysis, so was not analyzed at the final analysis; Test type: Superiority; p = 1.0, Log Rank; The log rank test was stratified by the factors provided at randomization; Hazard Ratio (HR) = 0.972, 98% CI 2-sided [0.726 to 1.00] — The hazard ratio estimate compares Cediranib to chemotherapy. If Cediranib is superior, the hazard ratio is <1.0

3. Primary Outcome: Overall Survival (OS) (Phase III Only)
Description: Overall survival will be evaluated. To allow for better understanding of time to subsequent therapy and OS, patients on experimental study drug(s) or standard chemotherapy arm will be followed after progression, with data capture to include the date of initiation of the subsequent therapy, detailed information on the type of subsequent therapy received, and time to progression on the subsequent therapy.
Time Frame: Time from study enrollment to death due to any cause, assessed up to 5 years
Population: All randomized subjects in Arms I - VII (excluding Arm IV).
  Arm 4 (Olaparib alone) was not continued in the Phase III part for its lack of efficacy after the completion of the Phase II portion. No further analyses were performed or reported for this arm.
  Twenty Japanese patients who were enrolled after the primary Phase III endpoint was reached were not included in the analysis for overall survival.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm V: (Arm I Regimen: JP Patients Enrolled After P3 Cutoff): Patients undergo physician's choice of standard of care chemotherapy, comprising either paclitaxel intravenously (IV) over 60 minutes on days 1, 8, 15, and 22 every 28 days (Regimen I); pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1 every 28 days (Regimen II); or topotecan hydrochloride IV over 30 minutes on days 1, 8, and 15 every 28 days or days 1-5 every 21 days (Regimen III). Treatment continues in the absence of disease progression or unacceptable toxicity. No modification of the assigned regimens, such as additional drugs (gemcitabine, or bevacizumab) is allowed. Patients also undergo computed tomography (CT) and magnetic resonance imaging (MRI) throughout the study. (12/05/2016) Patients enrolled from Japan after the Phase III cutoff.
Arm/Group | Arm I (Reference Regimen) | Arm II (Cediranib Maleate, Olaparib) | Arm III (Cediranib Maleate) | Arm V: (Arm I Regimen: JP Patients Enrolled After P3 Cutoff) | Arm VI: (Arm II Regimen: JP Patients Enrolled After P3 Cutoff) | Arm VII: (Arm III Regimen: JP Patients Enrolled After P3 Cutoff)
Number analyzed (Participants) | 173 | 167 | 170 | 5 | 8 | 7
months | 13.6 [11.6 to 15.8] | 12.8 [10.1 to 15.3] | 10.5 [9.1 to 12.3] | 14.9 [10.4 to NA] — The sample size is not sufficient for the estimation of the upper bound of the CI. | 18.0 [2.8 to NA] — The sample size is not sufficient for the estimation of the upper bound of the CI. | 5.8 [3.6 to 17.5]
Statistical Analysis 1: Comparison: Arm I (Reference Regimen) vs Arm II (Cediranib Maleate, Olaparib); Arm IV was suspended for futility at the end of Phase 2 analysis, so was not analyzed at the final analysis; Test type: Superiority; No p-values are provided because testing each of these null hypotheses was conditioned on first rejecting hypothesis concerning PFS; Hazard Ratio (HR) = 1.027, 98% CI 2-sided [0.771 to 1.368] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm I (Reference Regimen) vs Arm III (Cediranib Maleate); Arm IV was suspended for futility at the end of Phase 2 analysis, so was not analyzed at the final analysis; Test type: Other — No p-values are provided because testing each of these null hypotheses was conditioned on first rejecting hypothesis concerning PFS; [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 1.060, 98% CI 2-sided [0.795 to 1.413] — The hazard ratio estimate compares Cediranib to chemotherapy. If Cediranib is superior, the hazard ratio is <1.0

4. Secondary Outcome: Objective Response Rate (Complete Response and Partial Response) (Phase II Only)
Description: The Response Rates were estimated as the binomial proportion of patients with Best Overall Response of Complete or Partial response according to RECIST 1.1 criteria.
  A Complete response (CR) is defined as the complete disappearance of all target lesions, while a Partial response (PR) is defined as at least a 30% decrease in the sum of the longest diameters of target lesions compared to the baseline measurement; essentially, the tumor shrinks significantly but does not completely disappear. Overall response (OR) = CR + PR.
Time Frame: Up to 5 years
Population: Patients randomized at phase II and with measurable disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Reference Regimen) | Arm II (Cediranib Maleate, Olaparib) | Arm III (Cediranib Maleate) | Arm IV (Olaparib) (Phase II Only)
Number analyzed (Participants) | 46 | 53 | 51 | 49
Participants | 4 | 17 | 9 | 3

5. Secondary Outcome: Objective Response Rate (Complete Response and Partial Response for Phase III Only)
Description: as for outcome 4
Time Frame: Up to 5 years
Population: Patients with measurable disease in Arms I - VII (excluding Arm IV).
  Arm 4 (Olaparib alone) was not continued in the Phase III part for its lack of efficacy after the completion of the Phase II portion. No further analyses were performed or reported for this arm.
  Twenty Japanese patients who were enrolled after the primary Phase III endpoint was reached were not included in the analysis of overall response rates.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Reference Regimen) | Arm II (Cediranib Maleate, Olaparib) | Arm III (Cediranib Maleate) | Arm V: (Arm I Regimen: JP Patients Enrolled After P3 Cutoff) | Arm VI: (Arm II Regimen: JP Patients Enrolled After P3 Cutoff) | Arm VII: (Arm III Regimen: JP Patients Enrolled After P3 Cutoff)
Number analyzed (Participants) | 93 | 90 | 96 | 5 | 8 | 7
Participants | 15 | 32 | 23 | 0 | 3 | 2

6. Secondary Outcome: Incidence of Grade 3 (or Higher) Adverse Events
Description: Adverse events will be categorized by CTCAE V4.0. This outcome will report the count of participants who experienced a grade 3 (or higher) adverse event.
Time Frame: Up to 5 years
Population: Randomized and treated patients in Arms I - VII.
  Arm 4 (Olaparib alone) was not continued in the Phase III part for its lack of efficacy after the completion of the Phase II portion. No further analyses were performed or reported for this arm.
  Twenty Japanese patients who were enrolled after the primary Phase III endpoint was reached were not included in the analysis of adverse events.
Measure: Count of Participants; unit: Participants
Groups:
- Arm IV (Olaparib) (Phase II Only): Patients receive olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI throughout the study. (In July 2018, the Data Monitoring Committee voted to exclude the olaparib alone regimen).
  Computed Tomography: Undergo CT
Arm/Group | Arm I (Reference Regimen) | Arm II (Cediranib Maleate, Olaparib) | Arm III (Cediranib Maleate) | Arm IV (Olaparib) (Phase II Only) | Arm V: (Arm I Regimen: JP Patients Enrolled After P3 Cutoff) | Arm VI: (Arm II Regimen: JP Patients Enrolled After P3 Cutoff) | Arm VII: (Arm III Regimen: JP Patients Enrolled After P3 Cutoff)
Number analyzed (Participants) | 156 | 163 | 162 | 49 | 5 | 7 | 7
Participants | 88 | 129 | 126 | 24 | 3 | 4 | 5

7. Other Pre Specified Outcome: Patient-reported Scores of Disease-related Symptoms
Description: Measured by the 9-item Disease Related Symptoms (DRS-9) subscale of the National Comprehensive Cancer Network (NCCN)-Functional Assessment of Cancer Therapy (FACT) Ovarian Symptom Index (NFOSI-18).
Time Frame: Up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Gene Mutations Assessed BROCA-HR
Description: A single proportional hazards model will be used to estimate the treatment hazard ratios (and variances) for each of the experimental treatments selected for phase III evaluation relative to the reference treatment (chemotherapy) group. The model will include adjustments for prior platinum-free interval, prior bevacizumab treatment, age at study enrollment, randomly assigned study treatment and BROCA-HR status. The estimated hazard ratio(s) for BROCA-HR and the corresponding confidence intervals will be depicted with a forest plot, and assessed for qualitative interaction(s).
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Circulating Endothelial Cell Levels
Description: A proportional hazards model will be used to assess a linear association between the change in circulating endothelial cell values and the log relative hazard of death within each treatment group. Sensitivity analyses will include known prognostic factors in the model. A plot of the martingale residuals or estimated relative hazards by change in circulating endothelial cell quintiles will be used to qualitatively assess the assumption of a linear relationship between the change in circulating endothelial cell values and the log relative hazard.
Time Frame: Baseline up to 5 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Biomarkers in Plasma Angiome
Description: A proportional hazards model will be used to assess whether the pretreatment values of any of these analytes have a prognostic association with overall survival. The model will include clinical covariates: age, performance status, and the randomly assigned study treatment. Proportional hazards models will be used to assess the relationship between patients' analyte values and log hazard. A proportional hazards model will be used to assess the potential predictive associations between analytes, treatment and survival.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Adverse events will be categorized by CTCAE V5.0. Adverse events will be summarized by treatment group, system organ class, and preferred term.
  All-cause mortality population is related to OS and therefore is all randomized patients (ITT) but the reporting population for AE (AE and SAE) is the safety population and is only the set of patients that received treatment (the purpose is to identify adverse events that are potentially related to treatment).
Arm/Group | Arm I (Reference Regimen) | Arm II (Cediranib Maleate, Olaparib) | Arm III (Cediranib Maleate) | Arm IV (Olaparib) (Phase II Only) | Arm V (Arm I Regimen: JP Patients Enrolled After P3 Cutoff) | Arm VI: (Arm II Regimen: JP Patients Enrolled After P3 Cutoff) | Arm VII: (Arm III Regimen: JP Patients Enrolled After P3 Cutoff)
All-Cause Mortality (participants affected / at risk) | 137/173 | 145/167 | 143/170 | 45/52 | 2/5 | 5/8 | 6/7
Serious Adverse Events (participants affected / at risk) | 12/156 | 21/163 | 19/162 | 14/49 | 0/5 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 151/156 | 162/163 | 162/162 | 46/49 | 5/5 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Reference Regimen) (N=156) | Arm II (Cediranib Maleate, Olaparib) (N=163) | Arm III (Cediranib Maleate) (N=162) | Arm IV (Olaparib) (Phase II Only) (N=49) | Arm V (Arm I Regimen: JP Patients Enrolled After P3 Cutoff) (N=5) | Arm VI: (Arm II Regimen: JP Patients Enrolled After P3 Cutoff) (N=7) | Arm VII: (Arm III Regimen: JP Patients Enrolled After P3 Cutoff) (N=7)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 5 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 4 | 2 | 0 | 0 | 0
Anal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Colonic perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ileal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 3 | 3 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 3 | 2 | 1 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 4 | 3 | 0 | 0 | 0
Death NOS (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 3 | 2 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peritoneal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
INR increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Weight loss (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0
Visceral arterial ischemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Reference Regimen) (N=156) | Arm II (Cediranib Maleate, Olaparib) (N=163) | Arm III (Cediranib Maleate) (N=162) | Arm IV (Olaparib) (Phase II Only) (N=49) | Arm V (Arm I Regimen: JP Patients Enrolled After P3 Cutoff) (N=5) | Arm VI: (Arm II Regimen: JP Patients Enrolled After P3 Cutoff) (N=7) | Arm VII: (Arm III Regimen: JP Patients Enrolled After P3 Cutoff) (N=7)
Anemia (Blood and lymphatic system disorders) | 65 | 35 | 22 | 27 | 1 | 1 | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 5 | 4 | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Conduction disorder (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Heart failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 3 | 3 | 3 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary valve disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 5 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 7 | 7 | 9 | 0 | 0 | 0 | 0
Tricuspid valve disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 5 | 3 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 3 | 2 | 1 | 0 | 0 | 0
Endocrine disorders - Other, specify (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 11 | 14 | 0 | 0 | 0 | 0
Hypoparathyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 44 | 55 | 1 | 0 | 3 | 3
Blurred vision (Eye disorders) | 2 | 7 | 10 | 2 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 4 | 3 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flashing lights (Eye disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Floaters (Eye disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal vascular disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitreous hemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Watering eyes (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 8 | 12 | 6 | 3 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 47 | 61 | 65 | 15 | 0 | 1 | 1
Anal mucositis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 12 | 6 | 4 | 3 | 0 | 0 | 0
Bloating (Gastrointestinal disorders) | 14 | 12 | 15 | 2 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colonic hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 4 | 5 | 2 | 0 | 0 | 0 | 0
Colonic perforation (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 44 | 54 | 33 | 9 | 0 | 1 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 34 | 122 | 124 | 13 | 1 | 5 | 5
Dry mouth (Gastrointestinal disorders) | 2 | 20 | 25 | 1 | 0 | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 18 | 18 | 11 | 2 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 7 | 8 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 0 | 1 | 0
Esophageal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Esophageal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Fecal incontinence (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 4 | 5 | 5 | 0 | 0 | 0 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 16 | 13 | 11 | 2 | 0 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 6 | 9 | 6 | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Gastroparesis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 10 | 3 | 0 | 0 | 0 | 0
Ileal obstruction (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 2 | 1 | 3 | 2 | 0 | 1 | 1
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 41 | 42 | 57 | 3 | 1 | 2 | 3
Nausea (Gastrointestinal disorders) | 77 | 111 | 91 | 34 | 1 | 2 | 2
Obstruction gastric (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Oral dysesthesia (Gastrointestinal disorders) | 0 | 5 | 5 | 0 | 0 | 0 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 2 | 8 | 8 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 6 | 0 | 5 | 1 | 0 | 0 | 0
Rectal mucositis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal pain (Gastrointestinal disorders) | 2 | 1 | 4 | 0 | 0 | 0 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 14 | 12 | 13 | 3 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 3 | 2 | 2 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 32 | 78 | 59 | 16 | 1 | 0 | 1
Chills (General disorders) | 1 | 8 | 4 | 2 | 0 | 0 | 0
Death NOS (General disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0
Edema limbs (General disorders) | 20 | 19 | 20 | 7 | 0 | 0 | 0
Edema trunk (General disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 84 | 124 | 104 | 28 | 0 | 1 | 0
Fever (General disorders) | 9 | 6 | 8 | 1 | 0 | 0 | 0
Flu like symptoms (General disorders) | 3 | 6 | 3 | 2 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 3 | 3 | 0 | 0 | 0 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 3 | 5 | 4 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (General disorders) | 6 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0
Injection site reaction (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Irritability (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localized edema (General disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 3 | 1 | 1 | 0 | 3 | 4
Non-cardiac chest pain (General disorders) | 4 | 5 | 4 | 1 | 0 | 0 | 0
Pain (General disorders) | 16 | 14 | 13 | 10 | 0 | 0 | 0
Sudden death NOS (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 1
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 3 | 5 | 3 | 0 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bladder infection (Infections and infestations) | 1 | 2 | 2 | 0 | 0 | 0 | 0
Bronchial infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Gum infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 10 | 13 | 8 | 0 | 0 | 0 | 0
Lip infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 4 | 3 | 2 | 0 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Papulopustular rash (Infections and infestations) | 4 | 3 | 0 | 0 | 0 | 0 | 0
Peritoneal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 5 | 6 | 3 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 3 | 3 | 3 | 2 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 4 | 7 | 2 | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 17 | 26 | 25 | 3 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vulval infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 3 | 5 | 4 | 0 | 0 | 0 | 1
Burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 8 | 6 | 1 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 4 | 0 | 0 | 0 | 0 | 0
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prolapse of intestinal stoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 13 | 16 | 31 | 3 | 1 | 3 | 2
Alkaline phosphatase increased (Investigations) | 17 | 20 | 24 | 5 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 12 | 19 | 29 | 3 | 1 | 2 | 1
Blood bilirubin increased (Investigations) | 3 | 7 | 13 | 2 | 0 | 0 | 0
CPK increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac troponin I increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cholesterol high (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 11 | 31 | 31 | 8 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
GGT increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hemoglobin increased (Investigations) | 0 | 7 | 9 | 0 | 0 | 0 | 0
INR increased (Investigations) | 2 | 1 | 3 | 0 | 0 | 0 | 0
Investigations - Other, specify (Investigations) | 1 | 6 | 9 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 23 | 14 | 8 | 6 | 0 | 0 | 0
Lymphocyte count increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 54 | 23 | 12 | 4 | 3 | 2 | 1
Platelet count decreased (Investigations) | 24 | 34 | 30 | 6 | 0 | 3 | 3
Weight gain (Investigations) | 3 | 1 | 0 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 19 | 45 | 43 | 6 | 0 | 0 | 3
White blood cell decreased (Investigations) | 47 | 20 | 9 | 8 | 2 | 3 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 38 | 64 | 68 | 21 | 1 | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 6 | 25 | 30 | 3 | 0 | 0 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 6 | 7 | 3 | 3 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 24 | 26 | 16 | 3 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 6 | 10 | 3 | 0 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 1 | 0 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 19 | 19 | 23 | 6 | 0 | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 13 | 8 | 10 | 4 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 2 | 2 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 22 | 24 | 30 | 4 | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 10 | 14 | 21 | 5 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 16 | 27 | 26 | 10 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 0 | 3 | 2 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 16 | 12 | 2 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 5 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 16 | 24 | 4 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 0 | 0 | 1 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 3 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 5 | 1 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 | 19 | 23 | 3 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 0 | 0 | 0 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 10 | 5 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 15 | 23 | 6 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 4 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 21 | 13 | 4 | 0 | 0 | 0
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 4 | 1 | 0 | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Concentration impairment (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 9 | 26 | 27 | 3 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 0
Dysesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 9 | 19 | 20 | 4 | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 15 | 50 | 53 | 8 | 0 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 5 | 1 | 0 | 0 | 0 | 0
Myelitis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 4 | 2 | 2 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 23 | 21 | 21 | 4 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 0
Sinus pain (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stroke (Nervous system disorders) | 0 | 4 | 4 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 0
Transient ischemic attacks (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 4 | 2 | 3 | 0 | 0 | 0 | 0
Vasovagal reaction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 8 | 21 | 7 | 4 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 7 | 7 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 10 | 9 | 9 | 3 | 0 | 0 | 0
Hallucinations (Psychiatric disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 11 | 12 | 13 | 5 | 1 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Personality change (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 4 | 12 | 0 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 3 | 0 | 4 | 2 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 3 | 6 | 7 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 8 | 21 | 19 | 3 | 1 | 2 | 4
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 | 2 | 3 | 0 | 0 | 0 | 0
Renal calculi (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 7 | 4 | 5 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 7 | 3 | 2 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 2 | 2 | 2 | 1 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 5 | 5 | 4 | 0 | 0 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 3 | 2 | 1 | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 5 | 2 | 3 | 0 | 0 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Uterine hemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 3 | 4 | 2 | 3 | 0 | 0 | 0
Vaginal dryness (Reproductive system and breast disorders) | 4 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 | 3 | 3 | 2 | 0 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 5 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 19 | 27 | 5 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 38 | 47 | 40 | 15 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 9 | 5 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 | 18 | 28 | 0 | 0 | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 5 | 1 | 0 | 0 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 7 | 2 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 | 8 | 12 | 0 | 0 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 18 | 18 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 8 | 2 | 2 | 0 | 1 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 9 | 6 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 3 | 3 | 1 | 0 | 0 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 0 | 0 | 0 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 26 | 9 | 14 | 0 | 0 | 3 | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 8 | 3 | 2 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 2 | 5 | 1 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 30 | 13 | 12 | 6 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6 | 11 | 6 | 1 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 10 | 0 | 0 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2 | 3 | 2 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0
Hematoma (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 4 | 6 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 21 | 106 | 128 | 5 | 0 | 2 | 6
Hypotension (Vascular disorders) | 5 | 9 | 15 | 0 | 0 | 0 | 0
Lymphedema (Vascular disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 12 | 9 | 12 | 2 | 0 | 0 | 0
Vascular disorders - Other, specify (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visceral arterial ischemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT02502266/Prot_SAP_000.pdf